CLINICAL TRIAL: NCT03463850
Title: Multidimensional Analysis of Bone Micro-Architecture as a Clinical Biomarker for Image-Based Quantitative Fracture Risk Estimation.
Brief Title: Analysis of Bone Micro-Architecture as a Clinical Biomarker for Image-Based Fracture Risk Estimation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Kent Ogden, PhD, State University of New York - Upstate Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SUNYUMU 713378
Record Dates: First submitted 2016-07-14; First posted 2018-03-13 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Non-fracture (Experimental): subjects without a lumbar fracture will have a Dexa scan and Dual Energy CT (DECT) scan for observation/evaluation
  Interventions: Radiation: Dual Energy CT (DECT); Radiation: DEXA
- Fracture (Experimental): subjects with one or more lumbar fractures will have a Dexa scan andDual Energy CT (DECT) scan for observation/evaluation
  Interventions: Radiation: Dual Energy CT (DECT); Radiation: DEXA

INTERVENTIONS:
Radiation: Dual Energy CT (DECT) — Dual Energy CT (DECT)
Radiation: DEXA — Dual-energy x-ray absorptiometry for measurement of bone mineral density

SUMMARY:
Osteoporosis is a common disease among elderly people, which leads to an increased bone fracture risk. Bone fractures can greatly reduce quality of life and increase age-related problems including reduced life expectancy. In clinical practice, a bone mineral density (BMD) scan using dual-energy X-ray absorptiometry (DEXA) is used for diagnosing osteoporosis. However, DEXA does not always accurately predict who will develop fractures and who will not. This is because bone mineral density alone does not capture all of the factors that contribute to bone strength. One factor bone mineral density does not measure is trabecular microarchitecture of bone (structure of bone).

Our goal in this study is to use a specialized CT scan called Dual-Energy CT (DECT) to capture information about the trabecular (spongy) bone in the vertebra of the lower (lumbar) spine. Research has shown that this kind of information helps in predicting bone strength in bone specimens. The investigator will use this information to develop a method to more accurately predict which patients are likely to experience fractures of the lumbar vertebra. These are the most common type of fractures associated with osteoporosis.

The participant is being asked to participate in this research study because a physician is treating the participant for osteoporosis and the participant has met the initial criteria to participate in the study. Participation in this study involves having a DECT scan, as well as a DEXA scan if the participant has not had one recently (within two months).

Research studies include only those individuals who choose to take part. Please take time to make a decision. Please ask the study doctor or the study staff to explain any words or information that are not understood. The participant may also want to discuss it with family members, friends or other health care providers.

DETAILED DESCRIPTION:
Osteoporosis is a common disease among elderly people, the progression of which leads to an increased bone fracture risk, which can adversely affect quality of life and increase age-related morbidity/mortality. The National Osteoporosis Foundation forecast that by 2015, osteoporosis will be responsible for three million fractures resulting in $25.3 billion in healthcare costs. This highlights an urgent demand for methods to accurately predict osteoporotic fracture risk for clinical assessment and management of osteoporosis.

In clinical practice, dual-energy X-ray absorptiometry (DEXA) is the traditional and only method of diagnosing osteoporosis based on BMD measurements. However, DEXA has certain limitations, and a considerable overlap exists in BMD values between individuals who develop fractures and those who do not. This reflects that BMD does not capture all of the factors that contribute to bone strength. One such factor is trabecular microarchitecture of bone, well recognized in the definition of osteoporosis.

Ex vivo studies have demonstrated that trabecular bone microarchitecture constitutes an important component of bone strength, independent of BMD. However, trabecular microarchitecture is not considered in the evaluation of fracture risk in clinical practice. Several imaging techniques have been reviewed as potential candidates for clinical evaluation of trabecular bone microarchitecture. Technological improvements in high resolution X-ray imaging and MRI are providing increasingly accurate data on bone microarchitecture, but can be used only at peripheral sites (femur and forearm) and have not yet been incorporated into standardized clinical imaging protocols due to the lack of central site (lumbar spine) assessment, where osteoporotic fractures are most prevalent.

The current literature suggests a potential to increase the diagnostic accuracy of bone-strength prediction by incorporating advanced mathematical descriptors of bone structure. The project collaborators in Rochester have demonstrated that geometrical features characterizing the femoral trabecular compartment can complement conventional BMD measurements and improve bone strength prediction in ex vivo femur specimens. However, little effort has been made to actually utilize this complementary image information in clinical practice. This study should encourage the further development of these techniques and implementation into clinical practice.

Our goal is to start to bridge the gap between fundamental research on bone strength prediction and clinical management of osteoporosis, reflecting a translational research approach from "bench to bedside". To this end, a novel methodology will be evaluated by both a retrospective analysis and a prospective pilot study. The specific choice of using dual-energy CT (DECT) for the prospective pilot study is motivated by the potential to improve BMD measurement beyond what Quantitative CT (QCT) can, and it also allows for material decomposition into calcium and soft-tissue components, which has applications for other clinically relevant disease entities and will eventually result in the widespread availability of this relatively new technology.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or greater Caucasian female with confirmed osteoporosis via prior DEXA.
* Patients with known vertebral fractures (Genant Grade 2 or higher) and with no fractures (Genant Score <2) from prior DEXA/VFA analysis will be recruited.
* Patients with fractures must have at least one lumbar vertebral body with no fracture(s) (as seen on prior DEXA scan) for analysis.

Exclusion Criteria:

* Incidental finding to include pathology unrelated to osteoporosis that would directly affect bone architecture in the L spine (e.g. lytic bone lesions)
* Study DEXA scan reveals all lumbar vertebra have fractures (Genant >= 2)
* Orthopedic hardware in the lumbar spine region
* Unable to have a CT scan (e.g. too heavy for CT scan table, 660 lb. limit)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Development of a predictive software tool that will analyze dual-energy CT scans of the spine, and use the image information to estimate the probability of the patient to suffer an osteoporotic fracture. | 2 years
  Computer algorithms will be developed to differentiate patients with high risk of fracture from patients with low risk of fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Ogden, PhD, Principal Investigator — Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No